CLINICAL TRIAL: NCT03575975
Title: 3D X-ray Motion Analysis of Ankle-foot Motion After Total Ankle Replacement With Stryker STAR Implant
Brief Title: 3D X-ray Motion Analysis of Ankle-foot Motion After Total Ankle Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to lack of funding and unforeseen delays.
Sponsor: Georgia Institute of Technology (Other)
Collaborators: Emory University (Other); Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: Ankle XMA Project
Record Dates: First submitted 2018-06-19; First posted 2018-07-03 (Actual); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Ankle Arthroplasty; Prosthesis User; Joint Disease
Keywords: x-ray motion analysis; joint kinematics; functional range of motion
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Mobile-bearing ankle prosthesis user: Users of the Stryker Scandinavian Total Ankle Replacement (STAR) mobile-bearing prosthesis.
  Interventions: Device: Total Ankle Replacement Prosthesis
- Control: Healthy individual age- and gender-matched to a participant in the mobile-bearing prosthesis user group.
- Fixed-bearing ankle prosthesis user: Users of the INBONE II Total Ankle Replacement fixed-bearing prosthesis.
  Interventions: Device: Total Ankle Replacement Prosthesis

INTERVENTIONS:
Device: Total Ankle Replacement Prosthesis — Comparison of functional range of motion in users of Stryker Scandinavian Total Ankle Replacement (STAR) prosthesis to users of INBONE 2 Total Ankle Replacement prosthesis and to matched controls with intact ankle joints.
  Groups: Fixed-bearing ankle prosthesis user; Mobile-bearing ankle prosthesis user

SUMMARY:
Patients who have had a total ankle joint replacement surgery typically have limited movement in their ankles possibly due to the fact that commonly used ankle joint prosthetic devices only allow limited axes of motion.

This study will evaluate the ability of a Scandinavian Total Ankle Replacement (STAR) mobile-bearing prosthesis and INBONE 2 fixed-bearing prosthesis to restore triplanar motion in the tibiotalar (ankle) joint following a surgical arthroplasty (total joint replacement) procedure.

3D X-ray video motion analysis will be utilized to quantify range of motion measurements in two groups of ankle prosthesis users and a group of matched control participants.

DETAILED DESCRIPTION:
15 study participants will include those using a Stryker STAR prosthesis and a Wright Medical INBONE 2 prosthesis and a group of matched control subjects.

CT scans of lower limb anatomy (ankle-foot complex) will be obtained for all subjects to be converted into 3D bone surface models for use in the joint motion tracking software.

Each participant will participate in one day of data collection with an X-Ray Motion Analysis (XMA) system. High-speed biplanar XMA system will capture video images of the skeletal motions within the foot-ankle complex during normal movement. Subjects will walk and perform controlled movements in the capture volume within the XMA system.

Following data collection, the 3D bone surface models will be mapped to the sagittal (side view), coronal (front view), and axial (top view) plane skeletal motions demonstrated in the collected x-ray videos. Motion tracking data will then be used to accurately animate the 3D bone models to demonstrate the active range of ankle-foot joint motions during voluntary movement and gait.

Resulting range of motion measurements in dorsiflexion/plantarflexion, internal/external rotation, and inversion/eversion will be used to determine the extent to which normal motion in the ankle-foot complex has been restored in ankle prosthesis users.

ELIGIBILITY:
INCLUSION CRITERIA:

* Between 18 to 79 years of age.

Additional Inclusion criteria for mobile-bearing ankle prosthesis user group:

* Able to walk independently with their prosthesis at different self-selected speeds
* Implanted with Stryker Scandinavian Total Ankle Replacement (STAR) prosthesis at least one year prior to enrollment
* Pain free and radiologically normal
* Able to walk at preferred walking speed without an assistive device (e.g., cane, crutches, etc.)

Additional Inclusion criteria for control group:

* Within 3 years of age of one of the mobile-bearing ankle prosthesis user participants
* Same gender as the matched mobile-bearing ankle prosthesis user participant
* Not have a history of major musculoskeletal injuries
* Not have a history of major neuromuscular injuries

Additional Inclusion criteria for fixed-bearing ankle prosthesis users:

* Able to walk independently with their prosthesis at different self-selected speeds
* Implanted with INBONE 2 prosthesis at least one year prior to enrollment
* Pain free and radiologically normal
* Able to walk at preferred walking speed without an assistive device (cane, crutches, etc.)

EXCLUSION CRITERIA:

* Have dementia or an inability to give informed consent
* Have significant or chronic loss of hip or knee joint motion
* Have any subtalar or hindfoot fusion
* Have a history of dizziness and/or balance problems
* Have had any additional x-ray exposures in the past year that would put beyond the recommended annual dose for the study
* Are pregnant
* Exhibit evidence of polysubsidence (implant loosening)
* Exhibit evidence of a broken implant

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants meeting the eligibility criteria will be convenience-sampled from within the metro-Atlanta area. Eligible participants with either a STAR or INBONE 2 prosthesis will be identified from among clinical populations treated at the Emory University Hospital. Control group participants will be convenience-sampled from within the metro-Atlanta area.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hui Chang, PhD, Principal Investigator — Georgia Institute of Technology
Locations (1):
- Georgia Institute of Technology, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile-bearing Ankle Prosthesis User | Fixed-bearing Ankle Prosthesis User | Control
Started | 4 | 5 | 0
Completed | 3 | 5 | 0
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Control group participants were not enrolled due to early termination of the study.
Groups:
- Control: Healthy individual age- and gender-matched to a participant in the mobile-bearing prosthesis user group.
  No participants were enrolled due to premature study termination.
- Total: Total of all reporting groups
Arm/Group | Mobile-bearing Ankle Prosthesis User | Fixed-bearing Ankle Prosthesis User | Control | Total
Number analyzed (Participants) | 4 | 5 | 0 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (12.6) | 70.0 (7.5) |  | 69.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 |  | 6
  Male | 1 | 2 |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0
  Not Hispanic or Latino | 0 | 0 |  | 0
  Unknown or Not Reported | 4 | 5 |  | 9
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Tibiotalar Joint Angle Kinematics
Description: 3D range of motions of the tibiotalar (upper ankle) joint were recorded and analyzed using a biplanar x-ray motion analysis system. In particular, joint ranges of motion were tested in terms of dorsiflexion-plantarflexion, internal-external rotation, and inversion-eversion angles.
Time Frame: 1 year
Population: All participants who completed all aspects of the study protocol.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Mobile-bearing Ankle Prosthesis User | Fixed-bearing Ankle Prosthesis User
Number analyzed (Participants) | 3 | 5
degrees
  Dorsiflexion-Plantarflexion Angle | 6.74 (2.04) | 7.47 (4.05)
  Internal-External Rotation Angle | 6.28 (4.51) | 7.39 (3.63)
  Inversion-Eversion Angle | 5.68 (2.81) | 4.51 (2.13)

2. Secondary Outcome: Tibiotalar Joint Linear Translation Kinematics
Description: 3D range of linear motions of the tibiotalar (upper ankle) joint were recorded and analyzed using a biplanar x-ray motion analysis system. In particular, linear joint ranges of motion were tested in terms of the anteroposterior, mediolateral, and superior-inferior axes.
Time Frame: 1 year
Population: All participants who completed all aspects of the study protocol.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Mobile-bearing Ankle Prosthesis User | Fixed-bearing Ankle Prosthesis User
Number analyzed (Participants) | 3 | 5
mm
  Antero-posterior axis | 0.68 (1.44) | 1.47 (2.07)
  Medio-Lateral axis | 0.60 (1.41) | 1.13 (1.49)
  Superior-Inferior axis | 0.28 (0.30) | 0.20 (0.13)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected only during the period of study participation (typically less than 1 week).
Arm/Group | Mobile-bearing Ankle Prosthesis User | Fixed-bearing Ankle Prosthesis User
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5

LIMITATIONS AND CAVEATS:
An early termination of the study led to a smaller number of subjects enrolled/analyzed than originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT03575975/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT03575975/ICF_002.pdf